CLINICAL TRIAL: NCT01136473
Title: Mechanism of Aphakic and Pseudophakic Glaucoma in Pediatric Patients: Exploring the Pathophysiology Through Lens Epithelial Cell Culture and Isolation of Candidate Factors From Aqueous Humor
Brief Title: Mechanism of Aphakic and Pseudophakic Glaucoma in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Orna Geyer, Professor, Carmel Medical Center
Other Study IDs: CMC-10-0035-CTIL
Record Dates: First submitted 2010-05-27; First posted 2010-06-03 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Congenital Cataract; Aphakic or Pseudophakic Glaucoma
Keywords: congenital cataract; aphakic; pseudophakic glaucoma; pediatric patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- congenital cataract or aphakic glaucoma: children with congenital cataract or aphakic glaucoma

SUMMARY:
In cell cultures, lens epithelial cells and trabecular meshwork cells will be exposed to aqueous humor from pediatric eyes undergoing cataract removal surgery. Cytokine analysis of candidate factors will be performed before and after exposure to lens epithelial.

DETAILED DESCRIPTION:
Aqueous from the anterior chamber will be withdrawn before surgery. Then the lens capsule will be opened (capsulorhexis) and removed. The lens material will be removed. All 3 components will be sent to the lab.

Lens epithelial cells will be isolated and will be used in a co-culture setup with trabecular cells to investigate the interactions between lens cells and trabecular cells. Understanding the interaction between young and adult lens cells on trabecular cell will shed light on mechanism of infantile aphakic glaucoma.

Aqueous humor taken out before cataract surgery and before glaucoma operation of aphakic eyes will be used for analysis of growth factor and cytokines in the Aphakic eye using proteins membrane arrays. Eyes before cataract surgery will be used as controls. Such analysis will shed light on the possible factors affecting trabecular cells in aphakic eye.

ELIGIBILITY:
Inclusion Criteria:

* children with congenital cataract and are going to do removal surgery
* children with aphakic or pseudophakic glaucoma and are going to do glaucoma surgery
* both of parents are able to sign the INFORMED CONSENT FORM

Exclusion Criteria:

* patients with other eye diseases apart from congenital cataract(in children with congenital cataract) and aphakic or pseudophakic glaucoma (in children with aphakic or pseudophakic glaucoma)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children 0-18
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
cell culture | one year
  In cell cultures, lens epithelial cells and trabecular meshwork cells will be exposed to aqueous humor from pediatric eyes undergoing cataract removal surgery. Cytokine analysis of candidate factors will be performed before and after exposure to lens epithelial.

CONTACTS AND LOCATIONS:
Overall Officials: Orna Geyer, Prof, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel